CLINICAL TRIAL: NCT05305573
Title: A Phase IIb, Double-Blind, Randomized, Active Controlled, Multi-center, Non-inferiority Trial to Assess Immunogenicity and Safety of a Booster Vaccination With a Recombinant Protein RBD Fusion Dimer Candidate (PHH-1V) Against SARS-CoV-2, in Adults Fully Vaccinated With Adenovirus Vaccine Against COVID-19
Brief Title: Assessing the Immunogenicity and Safety of a HIPRA's Candidate Booster Vaccination in Adults Fully Vaccinated With Adenovirus Vaccine Against COVID-19.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hipra Scientific, S.L.U (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HIPRA HH-10
Record Dates: First submitted 2022-03-29; First posted 2022-03-31 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; SARS-CoV-2 Acute Respiratory Disease
MeSH Terms: conditions — COVID-19 | interventions — HIPRA COVID-19 vaccine; BNT162 Vaccine; Injections

STUDY DESIGN:
Intervention Model Description: This is a Phase IIb, double-blind, randomized, active controlled, multi-center, non-inferiority trial that aims to assess the immunogenicity and safety of a booster vaccination with a candidate vaccine.
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) Subjects and the clinical study team will remain blinded to treatment allocation.
  Clinical/pharmacy staff involved in study drug preparation will be aware of which vaccine the subject is receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Vaccine HIPRA 40 ug/dose (Experimental)
  Interventions: Biological: COVID-19 Vaccine HIPRA 40 ug/dose
- Comirnaty (Pfizer-BioNtech) 30 ug/dose concentrate for dispersion for injection (Active Comparator)
  Interventions: Biological: Comirnaty (Pfizer-BioNtech) 30 ug/dose concentrate for dispersion for injection

INTERVENTIONS:
Biological: COVID-19 Vaccine HIPRA 40 ug/dose — Subjects will receive one injection of COVID-19 Vaccine HIPRA (PHH-1V)
  Arms: COVID-19 Vaccine HIPRA 40 ug/dose
Biological: Comirnaty (Pfizer-BioNtech) 30 ug/dose concentrate for dispersion for injection — Subjects will receive one injection of Comirnaty Vaccine
  Arms: Comirnaty (Pfizer-BioNtech) 30 ug/dose concentrate for dispersion for injection

SUMMARY:
Phase IIb clinical trial to assess the Immunogenicity and Safety of a HIPRA's Candidate Booster vaccination (PHH-1V) in adults fully vaccinated with the adenovirus vaccine Vaxevria against COVID-19.

DETAILED DESCRIPTION:
The study population includes healthy adults aged above 18 years old who have received two doses of the Vaxevria vaccine, and are at least 91 days and less than 365 days after their second dose. Participants will be randomly assigned into two treatment arms. In each arm, volunteers will be randomized in a ratio Test vaccine:Comirnaty of 2:1. Each participant will receive one booster immunisation and will be followed for 6 months to evaluate immunogenicity response and assess the safety of the test vaccine in comparison to Comirnaty.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be considered eligible for the study:

1. Male or female, ≥ 18 years old at Day 0.
2. Participant must provide consent indicating that she or he understands the purpose and potential risks and is willing and able to participate in the study and comply with all the study requirements and procedures (scheduled visits, laboratory tests, complete diaries, etc).
3. Participant who has been vaccinated with two doses of Vaxzevria at least 91 days before Day 0 and a maximum of 365 days of the second dose.
4. Has a negative Rapid Antigen Test (RAT) at Day 0
5. Participants may have underlying illnesses if are stable and well-controlled according to the investigator judgment. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months prior to screening and for which neither a significant change in treatment or hospitalization for worsening is expected in the near future.
6. Participant agrees not to donate blood, blood products and bone marrow at least 12 weeks before and after vaccination.
7. Contraceptive use should be consistent with local regulation for participants in clinical trials.

   1. Female participants of childbearing potential [defined as any female who has experienced menarche and until becoming postmenopausal* (defined as having ≥ 12 months amenorrhea prior to screening without an alternative cause) unless is surgically sterile]: i. Have a negative pregnancy test on the day of vaccination. ii. Use of any acceptable contraceptive method that should be started at screening and until 8 weeks after vaccination except hormonal contraception. Acceptable contraceptive methods are:

1. Hormonal contraception (progestogen-only or combined): oral, injectable or transdermal (patch) at least 30 days before Day 0 and until 8 weeks after vaccination.

2. Intrauterine device. 3. Vasectomized partner (the vasectomized partner should be the sole partner for that participant).

4. Sexual abstinence **, as a form of contraception, is acceptable if in line with the participant's lifestyle.

5. Condom

b. Male participants: i. Vasectomized participants. ii. Refrain from donating sperm for at least 28 days after day 0. iii. Agree to use a male condom may be considered in women of childbearing potential partners, from screening and for at least 28 days after day 0. iv. Sexual abstinence**, as a form of contraception, is acceptable if in line with the participant's lifestyle.

* A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy.

** Sexual abstinence is considered an effective method only if defined as refraining from heterosexual intercourse from screening until 8 weeks after receiving the vaccine for female participants and from screening until 4 weeks for male participants. Periodic abstinence (e.g., calendar, ovulation) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study:

8. History of anaphylactic shock of any kind.

9. History of COVID-19 infection.

10. Participant received or plans to receive:

1. Live attenuated vaccines (licensed) within 4 weeks before or after receiving any study vaccine.
2. Other not live vaccines (licensed) within 14 days before and after receiving any study vaccine.

   11. Pregnancy or breast-feeding at screening or Day 0 (vaccination time-point) or willingness/intention to become pregnant during the study.

   Medical conditions:

   12. Participant has a clinically significant acute illness (this does not include minor self-limited illness such as mild diarrhoea) or fever (temperature ≥38º C (100.4ºF) at screening or within 48 hours prior to the planned vaccination (Day 0).

   13. Participant had a surgery requiring hospitalization (defined as inpatient stay for > 24 hours) before vaccination and he/she has not received the hospital discharge at day 0; or has a surgery requiring hospitalization planned within 12 weeks after study vaccine administration. Minor surgical procedures not requiring hospitalization are accepted.

   14. Participant has any active malignancy even if under treatment except for (at the discretion of the investigator): a. Non-melanoma adequately treated skin cancer without evidence of disease.

b. Adequately treated uterine cervical carcinoma in situ without evidence of disease.

c. Adequately treated anal carcinoma in situ without evidence of disease. d. Localized prostate cancer.

15. Participant has ongoing severe and non-stable psychiatric condition likely to affect participation in the study (e.g., ongoing and non-stable severe depression, recent suicidal ideation, severe eating disorder, psychosis).

16. Participant has a problematic or risk use of substances including alcohol (except tobacco) that can compromise the study follow-up. Problematic or risk use of psychoactive substances is understood as the one that causes evident damage, whether it is dependence or any other physical, psychological, or social problem or that carries a high risk of suffering these damages. The negative consequences that consumption causes to third parties could be included.

17. Participant has a bleeding disorder (e.g., factor deficiency, platelet disorder), blood dyscrasia, or continuous use of anticoagulants or has any condition that in the opinion of the investigator contraindicates intramuscular injections or frequent phlebotomy. The use of ≤ 325mg of aspirin or ≤ 75mg of clopidogrel per day as prophylaxis is permitted but not combined.

18. Participant has abnormal function of the immune system as in autoimmune diseases, asplenia, recurrent infections or congenital/acquired immunodeficiency. Participants under immune-modifying treatment for any cause. Permitted: participants with stable clinical conditions (e.g., autoimmune thyroiditis, celiac disease, type 1- diabetes) and participants living with HIV with CD4 T cell count ≥ 400 cells/mm3 under stable antiretroviral treatment with a fully suppressed viral load ≥ 1 year are permitted [one or two non-consecutives blips (HIV viral load ≤ 500 viral copies)].

19. Participants have clinically significant and unstable cardiovascular, respiratory, hepatic, neurological, gastrointestinal, renal, or any other medical disorder as judged by the investigator and defined as disease requiring hospitalization or addition of new treatments or major dose adjustments within 3 months before screening.

20. Chronic or recurrent administration (during at least 14 days) of systemic immunosuppressant medication (defined as given by oral or parenteral routes) within 12 weeks preceding the planned administration of study vaccine (Day 0). The use of an oral prednisone dose <10mg per day or equivalent, ocular, topical, inhaled and nasal corticoids are allowed.

21. Subject has received immunoglobulins and/or blood-derived products 12 weeks prior vaccination (Day 0) or expects to receive them during the study.

22. Participant received any immunotherapy (monoclonal antibodies, plasma) aimed to prevent or treat COVID-19 within 90 days preceding the planned administration of study vaccine. Monoclonal antibodies for other indications are allowed.

23. Participation in any research involving an investigational product (drug, biologic, device) within 12 weeks prior to vaccination and during the study.

24. Participant has donated ≥ 450ml of blood products within 12 weeks before screening.

25. Participant has any medical condition and/or finding that in the investigator opinion might increase participant risks, interfere with the study or impair interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Changes of the immunogenicity against Omicron strain at Day 14 | Day 14
  Neutralisation titre against Omicron strain measured as inhibitory concentration 50 (IC50) by a pseudovirion-based neutralisation assay (PBNA) and reported as reciprocal concentration for each individual sample and geometric mean titre (GMT) for descriptive statistics analysis at Baseline and at Day 14.
Safety and tolerability of PHH-1V as a booster dose | Day 7
  Number, percentage, and characteristics of solicited local and systemic reactions through Day 7 after vaccination.
Safety and tolerability of PHH-1V as a booster dose | Day 28
  Number, percentage, and characteristics of unsolicited local and systemic adverse events (AEs) through Day 28 after vaccination.
Safety and tolerability of PHH-1V as a booster dose | Day 182
  Number and percentage of serious adverse events (SAEs) through the study duration.
Safety and tolerability of PHH-1V as a booster dose | Day 182
  Number and percentage of adverse event of special interest (AESI) through the study duration.
Safety and tolerability of PHH-1V as a booster dose | Day 182
  Number and percentage of medically attended adverse events (MAAE) related to study vaccine through the study duration.
Safety and tolerability of PHH-1V as a booster dose | Days 14, 98 and 182
  Change from Baseline in safety laboratory parameters at Days 14, 98 and 182 after vaccination.

SECONDARY OUTCOMES:
Changes of the immunogenicity measured by PBNA against the Variants of Concern (VOC) | Days 14, 98 and 182
  Neutralisation titre against VOCs (Beta and Delta) measured as IC50 by PBNA and reported as reciprocal concentration for each individual sample and GMT for treatment group comparison at Baseline and Days 14, 98 and 182.
Changes of the immunogenicity measured by PBNA against Omicron | Day 14
  Geometric mean fold rise (GMFR) in neutralising antibodies titres against Omicron and VOCs (Beta and Delta) for treatment group comparison at Baseline and Day 14.
Changes of the immunogenicity measured by PBNA against Omicron | Days 98 and 182
  Neutralisation titre against Omicron measured as IC50 by PBNA and reported as reciprocal concentration for each individual sample and GMT for treatment group comparison at Days 98 and 182.
Changes of the immunogenicity measured by VNA against Omicron | Days 14, 98 and 182
  Neutralisation titre measured as inhibitory dilution 50 (ID50) against Omicron by a VNA and reported as reciprocal dilution for each individual sample, and GMT for treatment group comparison at Baseline and Day 14, 98 and 182. This analysis will only be performed in a subset of participants.
Changes of the immunogenicity measured by total antibody quantification using ECLIA | Days 14, 98 and 182
  Binding antibodies titre measured for each individual sample and GMT for treatment group comparison at Baseline and Days 14, 98 and 182.
Changes of the immunogenicity measured by total antibody quantification using ECLIA | Day 14
  Geometric mean fold rise (GMFR) in binding antibodies titre from Baseline and Days 14.
Changes of the immunogenicity measured by total antibody quantification using ECLIA | Days 14, 98 and 182
  Percentage of subjects that, after a booster dose, have a ≥4-fold change in binding antibodies titre from Baseline and Days 14, 98 and 182.

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital HM Modelo, A Coruña
  - Hospital Gregorio Marañón, Madrid
  - Hospital HM Sanchinarro, Madrid
  - Hospital HM Puerta del Sur, Móstoles
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital HM Rosaleda, Santiago de Compostela
  - Complejo Hospitalario Universitario de Vigo, Vigo

IPD SHARING:
Plan to Share IPD: No